CLINICAL TRIAL: NCT03569449
Title: Optimizing a Paraprofessional, Family Partner Navigation Model for Children
Brief Title: Family Partner Navigation for Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: H-37634; 1R01MH117123-01 (NIH)
Record Dates: First submitted 2018-06-15; First posted 2018-06-26 (Actual); Results first posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Health Behavior
Keywords: Family navigation; Family partners; Multiphase optimization strategy (MOST); Pediatric Symptom Checklist-17; Survey of Wellbeing of Young children (SWYC); Family Resource Scale; Federally qualified community health center
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Group 1- Goat (Experimental): Clinic-based visit, usual care, standard pediatric surveillance, and structured visits
  Interventions: Behavioral: Usual care; Behavioral: Clinic-based visits; Behavioral: Standard pediatric surveillance; Behavioral: Structured, schedule-based visits
- Group 2- Cow (Experimental): Clinic-based visit, usual care, enhanced pediatric surveillance, and structured visits
  Interventions: Behavioral: Usual care; Behavioral: Clinic-based visits; Behavioral: Structured, schedule-based visits; Behavioral: Enhanced pediatric surveillance
- Group 3- Horse (Experimental): Clinic-based visit, technology-enhanced care coordination, standard pediatric surveillance, and structured visits
  Interventions: Behavioral: Clinic-based visits; Behavioral: Standard pediatric surveillance; Behavioral: Structured, schedule-based visits; Behavioral: Technology enhanced care coordination
- Group 4- Pig (Experimental): Clinic-based visit, technology-enhanced care coordination, enhanced pediatric surveillance, and structured visits
  Interventions: Behavioral: Clinic-based visits; Behavioral: Structured, schedule-based visits; Behavioral: Enhanced pediatric surveillance; Behavioral: Technology enhanced care coordination
- Group 5- Sheep (Experimental): Clinic-based visit, usual care, standard pediatric surveillance, and individually-tailored visits
  Interventions: Behavioral: Usual care; Behavioral: Clinic-based visits; Behavioral: Standard pediatric surveillance; Behavioral: :Individually-tailored visits
- Group 6- Llama (Experimental): Clinic-based visit, usual care, enhanced pediatric surveillance, and individually-tailored visits
  Interventions: Behavioral: Usual care; Behavioral: Clinic-based visits; Behavioral: Enhanced pediatric surveillance; Behavioral: :Individually-tailored visits
- Group 7- Cat (Experimental): Clinic-based visit, technology-enhanced care coordination, standard pediatric surveillance, and individually-tailored visits
  Interventions: Behavioral: Clinic-based visits; Behavioral: Standard pediatric surveillance; Behavioral: Technology enhanced care coordination; Behavioral: :Individually-tailored visits
- Group 8- Dog (Experimental): Clinic-based visit, technology-enhanced care coordination, enhanced pediatric surveillance, and individually-tailored visits
  Interventions: Behavioral: Clinic-based visits; Behavioral: Enhanced pediatric surveillance; Behavioral: Technology enhanced care coordination; Behavioral: :Individually-tailored visits
- Group 9- Donkey (Experimental): Clinic and community visits, usual care coordination, standard pediatric surveillance, and structured visits
  Interventions: Behavioral: Usual care; Behavioral: Standard pediatric surveillance; Behavioral: Structured, schedule-based visits; Behavioral: Clinic-based visits and community visits
- Group 10- Bear (Experimental): Clinic and community visits, usual care coordination, enhanced pediatric surveillance, and structured visits
  Interventions: Behavioral: Usual care; Behavioral: Structured, schedule-based visits; Behavioral: Enhanced pediatric surveillance; Behavioral: Clinic-based visits and community visits
- Group 11- Tiger (Experimental): Clinic and community visits, technology enhanced care coordination, standard pediatric surveillance, and structured visits
  Interventions: Behavioral: Standard pediatric surveillance; Behavioral: Structured, schedule-based visits; Behavioral: Technology enhanced care coordination; Behavioral: Clinic-based visits and community visits
- Group 12- Lion (Experimental): Clinic and community visits, technology enhanced care coordination, enhanced pediatric surveillance, and structured visits
  Interventions: Behavioral: Structured, schedule-based visits; Behavioral: Enhanced pediatric surveillance; Behavioral: Technology enhanced care coordination; Behavioral: Clinic-based visits and community visits
- Group 13- Monkey (Experimental): Clinic and community visits, usual care coordination, standard pediatric surveillance, and individually-tailored visits
  Interventions: Behavioral: Usual care; Behavioral: Standard pediatric surveillance; Behavioral: :Individually-tailored visits; Behavioral: Clinic-based visits and community visits
- Group 14- Zebra (Experimental): Clinic and community visits, usual care coordination, enhanced pediatric surveillance, and individually-tailored visits
  Interventions: Behavioral: Usual care; Behavioral: Enhanced pediatric surveillance; Behavioral: :Individually-tailored visits; Behavioral: Clinic-based visits and community visits
- Group 15- Elephant (Experimental): Clinic and community visits, technology-enhanced care, standard pediatric surveillance, and individually-tailored visits
  Interventions: Behavioral: Standard pediatric surveillance; Behavioral: Technology enhanced care coordination; Behavioral: :Individually-tailored visits; Behavioral: Clinic-based visits and community visits
- Group 16- Giraffe (Experimental): Clinic and community visits, technology-enhanced care, enhanced pediatric surveillance, and individually-tailored visits
  Interventions: Behavioral: Enhanced pediatric surveillance; Behavioral: Technology enhanced care coordination; Behavioral: :Individually-tailored visits; Behavioral: Clinic-based visits and community visits

INTERVENTIONS:
Behavioral: Usual care — Family partners will keep records and communicate with families using standard information technology, including telephones, electronic medical records, and standard desktop software.
  Arms: Group 1- Goat; Group 10- Bear; Group 13- Monkey; Group 14- Zebra; Group 2- Cow; Group 5- Sheep; Group 6- Llama; Group 9- Donkey
Behavioral: Clinic-based visits — Family partners will be restricted to working at the primary care clinic - communication will be restricted to telephone, text, and clinic visits
  Arms: Group 1- Goat; Group 2- Cow; Group 3- Horse; Group 4- Pig; Group 5- Sheep; Group 6- Llama; Group 7- Cat; Group 8- Dog
Behavioral: Standard pediatric surveillance — Monitoring is determined by standard pediatric practice. Behavioral screening is usually done annually.
  Arms: Group 1- Goat; Group 11- Tiger; Group 13- Monkey; Group 15- Elephant; Group 3- Horse; Group 5- Sheep; Group 7- Cat; Group 9- Donkey
Behavioral: Structured, schedule-based visits — Family Partners will utilize a predetermined schedule of contacts with families
  Arms: Group 1- Goat; Group 10- Bear; Group 11- Tiger; Group 12- Lion; Group 2- Cow; Group 3- Horse; Group 4- Pig; Group 9- Donkey
Behavioral: Enhanced pediatric surveillance — In Massachusetts, behavioral screening is mandated at every pediatric visit, which for children in the target population (ages 3-12 years) is annually. With "enhanced monitoring," Family Partners will screen children using validated instruments quarterly and communicate results to the child's care team
  Arms: Group 10- Bear; Group 12- Lion; Group 14- Zebra; Group 16- Giraffe; Group 2- Cow; Group 4- Pig; Group 6- Llama; Group 8- Dog
Behavioral: Technology enhanced care coordination — Behavioral: technology enhanced care coordination FPs will also have access to Act.MD, a cloud-based care coordination and communication tool that offers the potential to improve communication with families, schools, and the primary care site through administration of online questions, videoconferencing, and common portals that can be used by parents and multiple providers (e.g., FP, pediatrician, teacher).
  Arms: Group 11- Tiger; Group 12- Lion; Group 15- Elephant; Group 16- Giraffe; Group 3- Horse; Group 4- Pig; Group 7- Cat; Group 8- Dog
Behavioral: :Individually-tailored visits — Family Partners will be able to meet with families on an as-needed basis, with no predetermined schedule of contacts
  Arms: Group 13- Monkey; Group 14- Zebra; Group 15- Elephant; Group 16- Giraffe; Group 5- Sheep; Group 6- Llama; Group 7- Cat; Group 8- Dog
Behavioral: Clinic-based visits and community visits — In clinic-based visits the Family Partner is restricted to working at the primary care clinic and communication is restricted to telephone, text, and clinic visits. However in conditions with clinic based and community visits, the Family Partners will be available to meet families in their home and community (as well as the clinic), and accompany families to community-based meetings at school or childcare.
  Arms: Group 10- Bear; Group 11- Tiger; Group 12- Lion; Group 13- Monkey; Group 14- Zebra; Group 15- Elephant; Group 16- Giraffe; Group 9- Donkey

SUMMARY:
Family Navigation (FN), an evidence-based care management strategy which is a promising intervention to help low income and minority families access timely mental health services. Despite significant evidence supporting the effectiveness of FN, concerns exist about the ability to disseminate FN to a broad population due to inefficiency and cost. The proposed study employs an innovative research methodology, the Multiphase Optimization STrategy (MOST), a framework for developing highly efficacious, efficient, scalable, and cost-effective interventions. The investigators will conduct a randomized experiment to assess the individual components of FN and identify which components and component levels have greatest effect on access to, and engagement in, diagnostic and treatment services for children with mental health disorders. This information then guides assembly of an optimized FN model that achieves the primary outcomes with least resource consumption and participant burden

DETAILED DESCRIPTION:
The goal of this study is to determine the optimal delivery of a Family Navigation (FN) model that increases engagement in services to address children's behavioral health. While there is strong evidence that navigation decreases barriers to care for low income and minority families, little is known about which specific components contribute to its efficacy. The investigators propose to use MOST, a pioneering, engineering-inspired framework, to assess the performance of individual intervention components and their interactions.

Delivery of FN will be systematically varied across four components, each of which is represented by a separate factor in the 2x2x2x2 factorial study design. Specifically, each family will be randomly assigned to one of two conditions within each of four factors or delivery strategies, defining sixteen separate experimental conditions. Strategies include: (A) technology-assisted delivery of care coordination using an innovative, web-based platform called Act.MD (compared to usual care); (B) clinic based FN + community-based (compared to clinic-based only); (C) enhanced symptom tracking using more frequent behavioral symptom tracking (compared to standard pediatric surveillance); and (d) individually-tailored visits (compared to a predetermined schedule of contacts). All children will be followed through the electronic health record (EHR) for 12 months, for outcomes in services access and symptom tracking.

The main effects will be estimated of the four experimental factors and their interactions on the study's primary outcome - family engagement in services to address their child's behavioral health. This information then guides assembly of an optimized FN model that achieves the primary outcomes with least resource consumption and participant burden.

Children will be enrolled if they have a positive behavioral health screen OR parent concern. A "watchful waiting" group for families of children with more mild symptoms and/or who do not choose to access child behavioral services at the time of the index visit with the Family Partner (FP) will be included. These families will be followed and child symptoms tracked at 3, 6, 9 and 12 months. If the watchful waiting children have an increase in symptom severity, and/or the family later desires services, they will have the opportunity to receive FN services and be randomized to a study condition.

ELIGIBILITY:
Inclusion Criteria:

All children who are 3-12 years old:

* who screen positive on the Survey of Wellbeing of Young Children (SWYC) (3-5 years) OR
* who screen positive on the Pediatric Symptom Checklist-17 (PSC-17) (6-12 years) OR
* whose parents indicate a behavioral health concern during any pediatric visit

Exclusion Criteria:

* Children who are already actively engaged in behavioral health specialty care services, defined as having had a behavioral health visit in the last 30 days, who do not require new additional services
* Children with active psychosis
* Children with safety concerns requiring emergency mental health services.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 312 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2024-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Feinberg, ScD, CPNP, Principal Investigator — Boston Medical Center and Boston University SPH
Locations (1):
- DotHouse Health, Dorchester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Broder-Fingert S, Kuhn J, Sheldrick RC, Chu A, Fortuna L, Jordan M, Rubin D, Feinberg E. Using the Multiphase Optimization Strategy (MOST) framework to test intervention delivery strategies: a study protocol. Trials. 2019 Dec 16;20(1):728. doi: 10.1186/s13063-019-3853-y. PMID 31842963

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The total enrolled refers to the number of dyads.
Pre-assignment Details: Both a parent or legal guardian and a child were included in the dyad. Dyads were randomized as a single unit to a condition.
Groups:
- Group 16- Giraffe: Clinic & community visits, technology-enhanced care, enhanced pediatric surveillance, & individually-tailored visits
Period: Overall Study
Arm/Group | Group 1- Goat | Group 2- Cow | Group 3- Horse | Group 4- Pig | Group 5- Sheep | Group 6- Llama | Group 7- Cat | Group 8- Dog | Group 9- Donkey | Group 10- Bear | Group 11- Tiger | Group 12- Lion | Group 13- Monkey | Group 14- Zebra | Group 15- Elephant | Group 16- Giraffe
Started | 20 (20 children and 20 parents/caregivers) | 24 (24 children and 24 parents/caregivers) | 18 (18 children and 18 parents/caregivers) | 19 (19 children and 19 parents/caregivers) | 21 (21 children and 21 parents/caregivers) | 17 (17 children and 17 parents/caregivers) | 19 (19 children and 19 parents/caregivers) | 20 (20 children and 20 parents/caregivers) | 19 (19 children and 19 parents/caregivers) | 21 (21 children and 21 parents/caregivers) | 20 (20 children and 20 parents/caregivers) | 19 (19 children and 19 parents/caregivers) | 19 (19 children and 19 parents/caregivers) | 18 (18 children and 18 parents/caregivers) | 19 (19 children and 19 parents/caregivers) | 19 (19 children and 19 parents/caregivers)
Completed | 20 | 22 | 18 | 17 | 20 | 17 | 19 | 20 | 19 | 21 | 20 | 19 | 19 | 18 | 18 | 19
Not Completed | 0 | 2 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: We did not collect data on parent/guardian age, race, ethnicity or gender therefore baseline characteristic data is based on the child of the dyad.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1- Goat | Group 2- Cow | Group 3- Horse | Group 4- Pig | Group 5- Sheep | Group 6- Llama | Group 7- Cat | Group 8- Dog | Group 9- Donkey | Group 10- Bear | Group 11- Tiger | Group 12- Lion | Group 13- Monkey | Group 14- Zebra | Group 15- Elephant | Group 16- Giraffe | Total
Number analyzed (Participants) | 20 | 24 | 18 | 19 | 21 | 17 | 19 | 20 | 19 | 21 | 20 | 19 | 19 | 18 | 19 | 19 | 312
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Child age
  years | 6.6 (3.0) | 7.0 (2.9) | 7.2 (3.0) | 7.1 (3.5) | 6.8 (3.5) | 7.4 (3.8) | 6.6 (2.9) | 6.6 (3.1) | 7.2 (2.8) | 6.7 (3.3) | 7.4 (3.1) | 6.8 (3.5) | 7.3 (3.3) | 7.4 (3.3) | 6.7 (3.1) | 7.3 (2.7) | 7.0 (3.1)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Child sex/gender
  Participants
    Male | 12 | 17 | 12 | 11 | 15 | 12 | 16 | 12 | 10 | 14 | 7 | 8 | 8 | 8 | 12 | 13 | 187
    Female | 8 | 7 | 6 | 8 | 6 | 4 | 3 | 8 | 9 | 6 | 11 | 11 | 11 | 10 | 7 | 6 | 121
    Refused to answer | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Child race/ethnicity
  Participants
    Black/African Am | 2 | 4 | 3 | 3 | 4 | 3 | 2 | 2 | 2 | 5 | 4 | 3 | 5 | 3 | 6 | 3 | 54
    Asian | 6 | 7 | 2 | 6 | 4 | 4 | 6 | 6 | 4 | 5 | 5 | 6 | 7 | 6 | 6 | 5 | 85
    White | 1 | 0 | 1 | 0 | 2 | 1 | 2 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 11
    Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3
    More than one race | 3 | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 14
    Other | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 11
    Hispanic | 8 | 12 | 9 | 9 | 10 | 7 | 7 | 8 | 9 | 9 | 9 | 8 | 6 | 8 | 7 | 8 | 134
Region of Enrollment [Number; unit: participants]
  United States | 20 | 24 | 18 | 19 | 21 | 17 | 19 | 20 | 19 | 21 | 20 | 19 | 19 | 18 | 19 | 19 | 312

OUTCOME MEASURES:

1. Primary Outcome: Goal Completion
Description: Successful behavioral health service goal completion obtained from the electronic health record including Family Partner's template documentation.
Time Frame: 6 months
Population: Data are available for all 312 dyads.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1- Goat | Group 2- Cow | Group 3- Horse | Group 4- Pig | Group 5- Sheep | Group 6- Llama | Group 7- Cat | Group 8- Dog | Group 9- Donkey | Group 10- Bear | Group 11- Tiger | Group 12- Lion | Group 13- Monkey | Group 14- Zebra | Group 15- Elephant | Group 16- Giraffe
Number analyzed (Participants) | 20 | 24 | 18 | 19 | 21 | 17 | 19 | 20 | 19 | 21 | 20 | 19 | 19 | 18 | 19 | 19
Participants | 9 | 9 | 7 | 9 | 7 | 6 | 2 | 4 | 7 | 4 | 6 | 6 | 10 | 3 | 5 | 6

2. Primary Outcome: Time to Goal Completion
Description: Time to goal completion obtained from the electronic health record including Family Partner's template documentation.
Time Frame: 18 months
Population: This outcome was calculated for dyads with successful goal completion. This measure examines goal completion up to 18 months from baseline.
Measure: Median (Full Range); unit: days
Arm/Group | Group 1- Goat | Group 2- Cow | Group 3- Horse | Group 4- Pig | Group 5- Sheep | Group 6- Llama | Group 7- Cat | Group 8- Dog | Group 9- Donkey | Group 10- Bear | Group 11- Tiger | Group 12- Lion | Group 13- Monkey | Group 14- Zebra | Group 15- Elephant | Group 16- Giraffe
Number analyzed (Participants) | 12 | 14 | 11 | 13 | 12 | 11 | 6 | 8 | 10 | 8 | 10 | 13 | 14 | 9 | 10 | 11
days
  number analyzed (Participants) | 12 | 14 | 10 | 13 | 12 | 11 | 6 | 8 | 10 | 8 | 9 | 12 | 14 | 8 | 10 | 11
  (all) | 168 [15 to 302] | 159.5 [0 to 212] | 179 [66 to 239] | 177 [28 to 428] | 184 [35 to 280] | 193 [40 to 374] | 218.5 [169 to 311] | 191 [59 to 287] | 179 [0 to 259] | 182 [36 to 240] | 190 [19 to 226] | 191 [127 to 390] | 173 [68 to 292] | 268.5 [136 to 502] | 190.5 [0 to 277] | 192.5 [25 to 307]

3. Secondary Outcome: Change in the Survey of Well-being of Young Children (SWYC)
Description: The Survey of Well-being of Young Children (SWYC) screens for cognitive, motor, language, and social-emotional development among children up to 5½ years of age. Behavioral symptoms were tracked using the SWYC's subscale called the Preschool Pediatric Symptom Checklist (PPSC). The PPSC is an 18-item questionnaire. The total score is summed and can range from 0 to 36. A PPSC total score of 9 or greater indicates that a child is "at risk". Change in the SWYC's PPSC subscale was calculated by finding the difference between the 6 month score and baseline. Participants with increased risk at 6-month is a change from a PPSC total score of below 9 at baseline (low risk) to a score of 9 or greater at 6-month (at risk). Decreased risk at 6-month is a change from a PPSC total score at or above 9 at baseline (at risk) to one below 9 at 6-month follow-up (low risk). No change is either both scores remained "at risk" or both scores remained "low risk".
Time Frame: baseline, 6 months
Population: This survey is appropriate for children 3-5 years of age therefore administered to a subset of children. In addition, the SWYC was part of the "enhanced" factor and therefore was only administered in 8 out of 16 conditions.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1- Goat | Group 2- Cow | Group 3- Horse | Group 4- Pig | Group 5- Sheep | Group 6- Llama | Group 7- Cat | Group 8- Dog | Group 9- Donkey | Group 10- Bear | Group 11- Tiger | Group 12- Lion | Group 13- Monkey | Group 14- Zebra | Group 15- Elephant | Group 16- Giraffe
Number analyzed (Participants) | 0 | 4 | 0 | 6 | 0 | 3 | 0 | 6 | 0 | 4 | 0 | 6 | 0 | 3 | 0 | 5
Participants
  Increased risk |  | 1 |  | 1 |  | 0 |  | 0 |  | 0 |  | 1 |  | 0 |  | 1
  Decreased risk |  | 0 |  | 1 |  | 2 |  | 2 |  | 0 |  | 1 |  | 1 |  | 1
  No change in risk |  | 3 |  | 4 |  | 1 |  | 4 |  | 4 |  | 4 |  | 2 |  | 3

4. Secondary Outcome: Change in Pediatric Symptom Checklist-17 (PSC-17)
Description: Scores from the Pediatric Symptom Checklist-17 (PSC-17) will be used to assess child symptoms. The PSC-17 is a 17-item psychosocial screen designed to recognize cognitive, emotional, and behavioral problems. A value of 0 is assigned to "Never", 1 to "Sometimes," and 2 to "Often". The total score is calculated as a sum each of the 17-item level scores, with a potential range of total scores of 0 to 34. A PSC-17 score of 15 or higher suggests the presence of significant behavioral or emotional problems or "at risk". Change in the Pediatric Symptom Checklist-17 (PSC-17) total score was calculated between the baseline and 6-month follow-up. Increased risk at 6-month is a change from a PSC-17 total score from below 15 at baseline to a score of 15 or greater at 6-month. Decreased risk at 6-month is a change from a PPSC total score at or above 15 at baseline to one below 15 at 6-month follow-up. No change is either both scores remained "at risk" or both scores remained "low risk".
Time Frame: baseline, 6 months
Population: This survey is appropriate for children 4-18 years old. It was administered to eligible children 5-12 years old in the study. In addition, the PSC-17 was part of the "enhanced" factor and therefore was only administered in 8 out of 16 conditions.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1- Goat | Group 2- Cow | Group 3- Horse | Group 4- Pig | Group 5- Sheep | Group 6- Llama | Group 7- Cat | Group 8- Dog | Group 9- Donkey | Group 10- Bear | Group 11- Tiger | Group 12- Lion | Group 13- Monkey | Group 14- Zebra | Group 15- Elephant | Group 16- Giraffe
Number analyzed (Participants) | 0 | 11 | 0 | 7 | 0 | 5 | 0 | 7 | 0 | 9 | 0 | 5 | 0 | 6 | 0 | 6
Participants
  Increased risk |  | 1 |  | 0 |  | 1 |  | 1 |  | 3 |  | 0 |  | 0 |  | 1
  Decreased risk |  | 1 |  | 2 |  | 0 |  | 0 |  | 1 |  | 0 |  | 1 |  | 2
  No change in risk |  | 9 |  | 5 |  | 4 |  | 6 |  | 5 |  | 5 |  | 5 |  | 3

5. Secondary Outcome: Satisfaction With Hospital Care Questionnaire (SHCQ)
Description: The Satisfaction with Hospital Care Questionnaire (SHCQ) addresses aspects of hospital care. Three subscales were used: Information (6 questions), Patient Autonomy (2 questions), and Emotional Support (3 questions). Each question is self rated on a scale of 1 to 10 where 1=poor and 10 = excellent. Total scores were summed across the three subscales. Total scores can range from 11 to 110. Higher scores suggest greater satisfaction with hospital care.
Time Frame: 6 months
Population: There were 75 parents who could not be reached through telephone calls for survey administration at the 6-month time frame.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1- Goat | Group 2- Cow | Group 3- Horse | Group 4- Pig | Group 5- Sheep | Group 6- Llama | Group 7- Cat | Group 8- Dog | Group 9- Donkey | Group 10- Bear | Group 11- Tiger | Group 12- Lion | Group 13- Monkey | Group 14- Zebra | Group 15- Elephant | Group 16- Giraffe
Number analyzed (Participants) | 17 | 16 | 16 | 15 | 16 | 11 | 17 | 17 | 13 | 15 | 16 | 14 | 14 | 12 | 14 | 14
score on a scale | 90.4 (18.5) | 91.6 (15.5) | 91.9 (12.0) | 96.4 (10.1) | 92.9 (13.1) | 89.3 (18.8) | 83.8 (19.0) | 92.5 (17.4) | 90.9 (20.5) | 83.6 (25.0) | 86.8 (21.2) | 89.7 (16.2) | 83.4 (17.2) | 94.1 (14.7) | 87.5 (22.9) | 87.3 (24.0)

6. Secondary Outcome: Interpersonal Relationship With Navigator (PSN-I)
Description: The Interpersonal Relationship with Navigator (PSN-I) tool is a validated 9-item scale with strong psychometric properties in samples of culturally diverse, underserved patients. For each item the participant can respond, "strongly disagree" =1, "disagree" =2, "are undecided"=3, "agree" =4, or "strongly agree" =5. Total scores are summed across the 9-items and can range from 9 to 45; higher scores indicate higher satisfaction with their interpersonal relationship with the patient navigator.
Time Frame: 6 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1- Goat | Group 2- Cow | Group 3- Horse | Group 4- Pig | Group 5- Sheep | Group 6- Llama | Group 7- Cat | Group 8- Dog | Group 9- Donkey | Group 10- Bear | Group 11- Tiger | Group 12- Lion | Group 13- Monkey | Group 14- Zebra | Group 15- Elephant | Group 16- Giraffe
Number analyzed (Participants) | 17 | 16 | 16 | 15 | 16 | 11 | 17 | 17 | 13 | 16 | 16 | 13 | 14 | 12 | 14 | 14
score on a scale | 31.4 (14.6) | 35.9 (11.1) | 30.6 (12.3) | 31.4 (13.3) | 30.4 (13.1) | 33.4 (13.3) | 32.1 (12.8) | 30.4 (10.8) | 30.5 (13.4) | 32.2 (11.5) | 33.1 (12.7) | 26.7 (12.9) | 32.9 (10.6) | 27.2 (12.9) | 34.3 (10.7) | 26.5 (11.4)

7. Secondary Outcome: Change in Family Resource Scale (FRS)
Description: The Family Resource Scale (FRS) is a 30-item scale assessing numerous family needs and factors: growth/support, health/necessities, physical necessities, physical shelter, intra-family support, communication/employment, child care, and personal resources. Each item is rated on a five-point scale ranging from "not-at-all-adequate" to "almost-always-adequate". Total scores were calculated by a sum across the 30-items. The minimum score is 30 and the maximum score is 150. Higher scores indicate more adequate levels of family resources.
  Change in score was calculated by taking the difference between total scores at baseline and 6 months. This was done by subtracting 6 month scores from baseline scores for each participant. Of note, a negative change value is due to a higher scores at baseline than at 6 months.
  The differences were averaged across the participants in each condition.
Time Frame: baseline, 6 months
Population: There were 75 parents who could not be reached through telephone calls for survey administration at the 6-month time frame. There were also 4 parents who completed less than 10% of the survey due to time constraints. Parents missing either a baseline or 6 month score could not be analyzed for a change in score.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1- Goat | Group 2- Cow | Group 3- Horse | Group 4- Pig | Group 5- Sheep | Group 6- Llama | Group 7- Cat | Group 8- Dog | Group 9- Donkey | Group 10- Bear | Group 11- Tiger | Group 12- Lion | Group 13- Monkey | Group 14- Zebra | Group 15- Elephant | Group 16- Giraffe
Number analyzed (Participants) | 17 | 16 | 16 | 15 | 16 | 10 | 17 | 16 | 13 | 16 | 15 | 14 | 13 | 12 | 14 | 13
score on a scale | 0.0 (0.6) | 0.3 (1.2) | 0.1 (0.4) | 0.1 (0.7) | 0.1 (9.7) | 0.0 (0.4) | 0.1 (0.7) | 0.6 (0.9) | 0.8 (0.9) | 0.2 (0.6) | 0.1 (0.5) | 0.2 (0.6) | 0.0 (0.7) | 0.0 (0.4) | 0.2 (0.6) | 0.5 (0.8)

8. Secondary Outcome: Change in Patient Health Questionnaire-2 (PHQ-2)
Description: The Patient Health Questionnaire-2 (PHQ-2) is a validated 2-question depression screening tool. PHQ-2 total score ranges from 0-6. The authors of the measure identified a score of 3 as the optimal cut-point when using the PHQ-2 to screen for depression. If the score is 3 or greater, major depressive disorder is likely.
  Change in score was calculated by taking the difference between total scores at baseline and 6 months. This was done by subtracting 6 month scores from baseline scores for each participant. Of note, a negative change value is due to a higher scores at baseline than at 6 months.
  The differences were averaged across the participants in each condition.
Time Frame: baseline, 6 months
Population: This survey was part of the "enhanced" factor and therefore was only administered to 8 out of 16 conditions. This survey was administered to the parents/guardians.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1- Goat | Group 2- Cow | Group 3- Horse | Group 4- Pig | Group 5- Sheep | Group 6- Llama | Group 7- Cat | Group 8- Dog | Group 9- Donkey | Group 10- Bear | Group 11- Tiger | Group 12- Lion | Group 13- Monkey | Group 14- Zebra | Group 15- Elephant | Group 16- Giraffe
Number analyzed (Participants) | 0 | 13 | 0 | 13 | 0 | 8 | 0 | 13 | 0 | 15 | 0 | 11 | 0 | 11 | 0 | 11
score on a scale |  | 0.2 (1.6) |  | -0.3 (0.5) |  | -1.1 (2.3) |  | -0.2 (2.4) |  | -0.5 (2.0) |  | -0.2 (1.6) |  | 0.4 (1.1) |  | 0.9 (2.0)

9. Secondary Outcome: Change in the Parental Attitudes Toward Psychological Services Inventory (PATPSI)
Description: The Parental Attitudes Toward Psychological Services Inventory (PATPSI) measure consists of 26 Likert-type items, assessing help-seeking attitudes, help-seeking intentions, and mental health stigma, and is scored on a Likert-type scale from 0 (strongly disagree) to 5 (strongly agree). Scores can range from 0 to 130. Higher scores are more favorable.
  Change in score was calculated by taking the difference between total scores at baseline and 6 months. This was done by subtracting 6 month scores from baseline scores for each participant. Of note, a negative change value is due to a higher scores at baseline than at 6 months.
  The differences were averaged across the participants in each condition.
Time Frame: baseline, 6 months
Population: There were 75 parents who could not be reached through telephone calls for survey administration at the 6-month time point. There were also 4 parents who completed less than 10% of the survey due to time constraints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1- Goat | Group 2- Cow | Group 3- Horse | Group 4- Pig | Group 5- Sheep | Group 6- Llama | Group 7- Cat | Group 8- Dog | Group 9- Donkey | Group 10- Bear | Group 11- Tiger | Group 12- Lion | Group 13- Monkey | Group 14- Zebra | Group 15- Elephant | Group 16- Giraffe
Number analyzed (Participants) | 17 | 16 | 15 | 15 | 16 | 10 | 17 | 17 | 13 | 15 | 14 | 14 | 14 | 12 | 14 | 14
score on a scale | -1.0 (5.0) | 1.2 (8.9) | 5.1 (5.9) | 0.5 (5.3) | 1.3 (6.3) | 0.3 (12.1) | -3.6 (6.1) | -1.3 (8.2) | -4.5 (7.9) | -0.2 (9.0) | -3.0 (8.0) | 1.2 (6.1) | -0.5 (8.1) | -2.3 (8.0) | -1.1 (6.5) | -2.2 (9.8)

ADVERSE EVENTS:
Time Frame: 18 months
Description: Adverse events were non-systematically assessed only for children. There were no adverse events reported.
Arm/Group | Group 1- Goat | Group 2- Cow | Group 3- Horse | Group 4- Pig | Group 5- Sheep | Group 6- Llama | Group 7- Cat | Group 8- Dog | Group 9- Donkey | Group 10- Bear | Group 11- Tiger | Group 12- Lion | Group 13- Monkey | Group 14- Zebra | Group 15- Elephant | Group 16- Giraffe
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/24 | 0/18 | 0/19 | 0/21 | 0/17 | 0/19 | 0/20 | 0/19 | 0/21 | 0/20 | 0/19 | 0/19 | 0/18 | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/24 | 0/18 | 0/19 | 0/21 | 0/17 | 0/19 | 0/20 | 0/19 | 0/21 | 0/20 | 0/19 | 0/19 | 0/18 | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/20 | 0/24 | 0/18 | 0/19 | 0/21 | 0/17 | 0/19 | 0/20 | 0/19 | 0/21 | 0/20 | 0/19 | 0/19 | 0/18 | 0/19 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-20): https://cdn.clinicaltrials.gov/large-docs/49/NCT03569449/Prot_SAP_001.pdf
  • Informed Consent Form (2023-03-03): https://cdn.clinicaltrials.gov/large-docs/49/NCT03569449/ICF_002.pdf